CLINICAL TRIAL: NCT04157504
Title: Clinical Factors Affecting Physical Functions in Lower Limb Burn Injury
Brief Title: Evaluation of Physical Functions in Lower Limb Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GO 17/419
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Burns; Burn Scar; Lower Limb Injury; Lower Limb Wound
Keywords: Burn Injury; Balance; Lower extremity function; burn scar
MeSH Terms: conditions — Burns; Leg Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group: Physical Function (Experimental): Forty patients with burn injury will be evaluated in this study. Lower extremity function, functional capacity, functional mobility, quality of life an scar tissue will be evaluated.
  Interventions: Other: Physical function assessment

INTERVENTIONS:
Other: Physical function assessment — Physical function assessment is a tool to evaluate mobility levels of patients

SUMMARY:
This study evaluates scar tissue, normal range of motion of lowr extremity joints, lower extremity functions, functional capacity, functional mobility, kinesiophobia and quality of life in lower limb burn injury.

DETAILED DESCRIPTION:
Patients with lower extremity burns experience problems with range of motion, muscle strength, balance and gait. These problems contribute to prolonged physical disability, return to work or deterioration of work capacity and thus lead to a negative impact on quality of life.

In addition to studies showing that quality of life and functions may be affected adversely after burn, there are studies showing that burn percentage, health-related quality of life and functional outcomes are affected. The aim of this study is to determine the effects of burn area (with or without joint), percentage of burns and hypertrophic scar on the patient's function in patients with lower extremity burns.

ELIGIBILITY:
Inclusion Criteria:

* Having a lower limb burns
* To be a volunteer to participate

Exclusion Criteria:

* orthopedic problems affecting gait and stance
* Having a neurological disorders
* Walking with assist device

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Function | 10 minutes
  The Lower extremity functional index is a questionnaire containing 25 items. The value of this questionnaire between 0 and 100. The higher value indicates worse physical function.
Nottingham health profile | 10 minutes
  Nottingham health profile is a questionnaire that evaluates quality of life. he lowest and highest scores that can be obtained from each sub-dimension of the scale are 0 and 100, respectively. 0 indicates the best health status while 100 indicates the worst health status.

SECONDARY OUTCOMES:
scar tissue assessment | 10 minutes
  The Patient and Observer Scar Assessment Scale consists of the total score of two numeric scales measured by the patient and a qualified observer. Each scale assesses the scar by six characteristics on 10-point scales with a 1 corresponding to normal skin and a 10 representing the worst imaginable condition for that characteristic. The Total Score of both scales is calculated by summing scores of the six items resulting in a range of 6 to 60.
Tampa kinesiophobia scale | 10 minutes
  This scale consists of a 17-item self-report questionnaire that measures the fear of re-injury because of movement. Items are scored on a 4-point Likert scale ranging from 1 "strongly disagree" to 4 "strongly agree". The total scores for scale range from 17 to 68. Maximum score means higher level of kinesiophobia.
Six minutes walk test | 10 minutes
  It was evaluated by six minutes walk test.The 6-min walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The distance will be recorded. The higher distance is indicated better exercise capacity.
Timed up and go test | 5 minutes
  Timed up and go test evaluates dynamic balance of participants. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.Timed up and go test measure is second. The lower values indicates the better balance

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No